CLINICAL TRIAL: NCT01444625
Title: Flavanols and Skin Photo Protection: a Double Blind Clinical Trial
Brief Title: Flavanols and Skin Photo Protection: a Clinical Trial
Acronym: CHOCOPO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Claudine Blanchet, Coordinator, Laval University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Callebaut-10151; Callebaut-10151 (Other: Barry Callebaut Canada Inc)
Record Dates: First submitted 2011-09-26; First posted 2011-10-03 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2012-05

CONDITIONS: Solar Skin Damage
Keywords: UV radiation; photoprotection; flavanols rich chocolate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dark chocolate (Experimental): Flavanol-rich chocolate
  Interventions: Other: Flavanol-rich chocolate
- Placebo chocolate (Placebo Comparator): Flavanol-free chocolate
  Interventions: Other: Flavanol-free chocolate

INTERVENTIONS:
Other: Flavanol-rich chocolate — High-flavanol chocolate, 12 weeks.
  Other Names: Experimental dark chocolate
  Arms: Dark chocolate
Other: Flavanol-free chocolate — Flavanol-free chocolate, 12 weeks
  Other Names: Placebo flavanol-free chocolate
  Arms: Placebo chocolate

SUMMARY:
As flavanols have antioxidants, anti-inflammatory and anti-DNA damaging effects and may increase microcirculation in skin, the purpose of the study is to investigate the chronic effect of flavanol-rich chocolate as an effective strategy to protect against the harmful effect of ultraviolet (UV) radiation.

DETAILED DESCRIPTION:
Recent data suggested that chronic ingestion of high flavanols cocoa might be a promising agent for dietary photo protection against UV light. Moreover, flavanols-rich cocoa intake has been shown to increase microcirculation in human skin.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking women between the ages of 20 and 65 years.
* Normal skin of type I and II as decried by Fitzpatrick classification.

Exclusion Criteria:

* Pregnancy and breast feeding.
* Photo sensibility: history of skin cancers, photosensitizing medication.
* Sun bed use or sunbathing in the previous 3 months.
* Use of supplements or natural health products (fish oils, coenzyme Q10, garlic, lycopene, beta carotene).
* Allergy or intolerance to nuts or chocolate.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2011-06; Primary Completion 2012-09 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change in Minimal erythema dose | within the first 12 weeks of chocolate intake and 3 weeks later after end of chocolate consumption

SECONDARY OUTCOMES:
Change in Skin elasticity | within the first 12 weeks of chocolate intake and 3 weeks later after end of chocolate consumption
Change in Skin moisture | within the first 12 weeks of chocolate intake and 3 weeks later after end of chocolate consumption
Change in levels of Vitamin D and polyphenols | within the first 12 weeks of chocolate intake and 3 weeks later after end of chocolate consumption

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Dodin, MD, Principal Investigator — Laval University
Locations (1):
- Laval university, Department of Medicine, Institut des nutraceutiques et des aliments fonctionnels., Québec, Quebec, Canada

REFERENCES:
- [Derived] Mogollon JA, Boivin C, Lemieux S, Blanchet C, Claveau J, Dodin S. Chocolate flavanols and skin photoprotection: a parallel, double-blind, randomized clinical trial. Nutr J. 2014 Jun 27;13:66. doi: 10.1186/1475-2891-13-66. PMID 24970388